CLINICAL TRIAL: NCT06392061
Title: Assessment of Medical and Nutritional Status Post-Probiotic Intake in Patients Diagnosed With Inflammatory Bowel Disease: A Randomized Clinical Trial
Brief Title: Effect of Probiotic Administration on Patients With Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Zahra SADEK, Associate Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LebaneseUni
Record Dates: First submitted 2024-04-18; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Quality of Life; Food Intolerance; Flare Up; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Food Intolerance; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Contains 4 strains of naturally-occurring bacteria including: Lactobacillus acidophilus, LA-5®, Bifidobacterium animalis, BB-12®, Streptococcus thermophiles, STY-31 and Lactobacillus delbrueckii subsp. Bulgaricus LBY-27 in concentration of 4.5 milliards CFU/capsule.
  Interventions: Dietary Supplement: Trilac
- Control (No Intervention): The patients will be asked to continue their usual lifestyle without change in their usual medication and nutritional intake.

INTERVENTIONS:
Dietary Supplement: Trilac — Trilac® is a dietary supplement developed by Surveal Pharma to support digestive health and overall well-being. This probiotic contains 4 strains of naturally-occurring bacteria including: Lactobacillus acidophilus, LA-5®, Bifidobacterium animalis, BB-12®, Streptococcus thermophiles, STY-31 and Lactobacillus delbrueckii subsp. Bulgaricus LBY-27 in concentration of 4.5 milliards CFU/capsule. Patients in the probiotic group will be instructed to take one tablet per day for a period of 8 weeks.
  Arms: Probiotic

SUMMARY:
The study is a single-center, randomized, single-blinded, controlled trial conducted at ZHUMC's endoscopy unit. It aims to assess the short-term effects of probiotic administration on disease course, quality of life, and nutritional status among patients diagnosed with inflammatory bowel disease (IBD), specifically ulcerative colitis (UC) and Crohn's disease (CD).

Patients with UC and CD will be recruited from the endoscopy unit's outpatients and divided into two groups: a control group and an intervention probiotic group. The intervention probiotic group will receive the probiotic intervention for 2 months. During the study period, two visits will be scheduled for all patients.

At each visit, medical and nutrition surveys will be filled out, and body composition measurements will be conducted. These assessments will help evaluate the impact of probiotic administration on the participants' disease progression, their quality of life, and their nutritional status.

Overall, the study aims to provide insights into the potential benefits of probiotic supplementation in managing IBD and improving the well-being of patients with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Lebanese outpatients with histological diagnosis of Crohn's disease or Ulcerative Colitis from at least 6 months prior to the trial.
* have stable inactive disease.
* have not used any probiotics within the two months before the investigation.

Exclusion Criteria:

* pregnant or lactating women
* patients who use probiotics within the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease course | 8 weeks
  Change in frequency of flares over 2 months
Disease course | 8 weeks
  Change in hospitalizations rates over 2 months
Nutrition Status | 8 weeks
  Change in macro- and micronutrient intake by administrating 24 h recall to be analysed by Nutritionist Pro Software

SECONDARY OUTCOMES:
Quality of Life Status | 8 weeks
  Change in quality-of-life score as per WHOQOL Bref

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hallal, Principal Investigator — Al Zahraa Hospital University Medical Center
Locations (1):
- zahra Sadek, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No